CLINICAL TRIAL: NCT04715048
Title: Split-Face Study Comparing OnabotulinumtoxinA (Botox) and PrabotulinumtoxinA (Jeuveau) in Treating Glabellar Lines
Brief Title: Split-Face Study Comparing Botox and Jeuveau in Treating Glabellar Lines
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Sandy Zhang-Nunes, Assistant Professor of Clinical Ophthalmology; Chief of Oculofacial Plastics Services, University of Southern California
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: HS-19-00455
Record Dates: First submitted 2021-01-10; First posted 2021-01-20 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Glabellar Frown Lines
Keywords: Botox, Jeuveau
MeSH Terms: interventions — prabotulinumtoxin A; onabotulinum toxin A; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The two different neurotoxins will be drawn into identical appearing syringes by an unblinded investigator. The injector will be a blinded investigator and will not know which syringe has which neurotoxin. There is no difference in appearance of the product when in a standardized syringe. The PI and co-investigator will be graders of these images and will be blinded during the grading process.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Onabotulinumtoxin A (Experimental): 8-10 units of Botox will be injected in the glabellar lines in one side of the face in 3 different locations. This injection will happen once.
  Interventions: Drug: Onabotulinum toxin A
- Prabotulinumtoxin A (Experimental): 8-10 units of Jeuveau will be injected in the glabellar lines in the other side of the face in 3 different locations. This injection will happen once.
  Interventions: Drug: PrabotulinumtoxinA

INTERVENTIONS:
Drug: PrabotulinumtoxinA — Glabellar line correction
  Other Names: Jeuveau
  Arms: Prabotulinumtoxin A
Drug: Onabotulinum toxin A — Glabellar line correction
  Other Names: Botox
  Arms: Onabotulinumtoxin A

SUMMARY:
The purpose of this study is to compare the efficacy and side effects of Botox and Jeuveau for glabellar lines.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients given consent will receive Botox on one side of their face and Jueveau on the other. A random number generator will generate a list of 20 combinations of "1,2" or "2,1". "1,2" means the Botox (onabotulinumtoxin A) will be placed on the right side and "2,1" means that the Botox will be placed on the left. The other side will be injected with PrabotulinumtoxinA. 8-10 units will be injected into the designated glabella in 3 sites.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Willingness to participate in the study and able to provide informed consent

Exclusion Criteria:

* Inability to follow up for study duration
* Prior neurotoxin injection in the last 4 months
* Prior surgery to the glabellar area
* Any planned aesthetic procedure to the glabellar area during the study period
* Cardiac Patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Movement on a 10 point Frown Movement Scale at 3 weeks | 3 weeks
  10-point scale created by the investigator assessing movement of glabellar lines. Possible scores range from 0 (no movement) to 10 (movement).

SECONDARY OUTCOMES:
Days to onset of neurotoxin | Up to 2-4 days
  # of days until neurotoxin begins decreasing movement on each side
Bruising from the injection on a scale of 1-10 | Up to 2-4 days
  Post injection bruising measured on a scale from 0 (no bruising) to 10 (most possible bruising) created by the investigator.
Pain from the injection on a scale of 1-10 | Up to 2-4 days
  Post injection pain will be measured on a scale from 0 (no pain) to 10 (most possible pain) created by the investigator.
Headache from the injection on a scale of 1-10 | Up to 2-4 days
  Post injection headache will be measured on a scale from 0 (no pain) to 10 (most possible pain) created by the investigator.
Movement on a 10 point Frown Movement Scale at 3 weeks | 3 weeks
  Patients grade their own movement of glabellar lines using a 10-point scale created by the investigator. Possible scores range from 0 (no movement) to 10 (movement).
Change in glabellar lines on the Merz Score (0-4) | At baseline and 3 weeks
  The Merz Score is a 5 point scale. The Merz Score will be used to grade glabellar lines at rest and frown at both baseline and the 3 week visit. Change will calculated from the 3 week visit compared to baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- USC Roski Eye Institute, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rzany BJ, Ascher B, Avelar RL, Bergdahl J, Bertucci V, Bodokh I, Carruthers JA, Cartier H, Delmar H, Denfeld R, Gross JE, Heckmann M, Heden P, Hilton S, Inglefield C, Ogilvie P, Sattler G, Sebastian M, Solish N, Swift A, Trevidic P. A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Single-Dose, Phase III, Non-Inferiority Study Comparing PrabotulinumtoxinA and OnabotulinumtoxinA for the Treatment of Moderate to Severe Glabellar Lines in Adult Patients. Aesthet Surg J. 2020 Mar 23;40(4):413-429. doi: 10.1093/asj/sjz110. PMID 30951166